CLINICAL TRIAL: NCT07266389
Title: Clinical Efficacy Evaluation of Supraglottic Airway Device SafeLM™ in Paediatric Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JEPUKM-JEP-2025-255
Record Dates: First submitted 2025-09-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia; Supraglottic Airway Efficiency; Paediatric Airway Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usage of SafeLM™ as the airway device (Experimental): SafeLM™ will be the airway device used for ventilation throughout the general anaesthesia period
  Interventions: Device: SafeLM™ as the airway management device during general anaesthesia

INTERVENTIONS:
Device: SafeLM™ as the airway management device during general anaesthesia — Appropriate size of SafeLM™ is selected for participants as manufacturer recommendation.
  Size 2 is for participants with body weight of 10-20 kg, recommended cuff volume to be inflated is 10 to 15 ml.
  Size 2.5 is for participants with body weight of 20-30 kg, recommended cuff volume to be inflated is 14 to 21 ml.
  Size 3 is for participants with body weight of 30-50 kg, recommended cuff volume to be inflated is 20 to 30 ml.
  Size 4 is for participants with body weight of 50-70 kg, recommended cuff volume to be inflated is 30 to 45 ml Size 5 is for participants with body weight of 70-100 kg, recommended cuff volume to be inflated is 40 to 60 ml.
  Under general anaesthesia, the device is held by the anaesthesiologist at the distal end while advancing the laryngeal mask by sliding down the palatopharyngeal curve along the midline in the mouth until the end of the mask reach the hypopharynx cavity and resistance is met, under direct real-time visualisation.

SUMMARY:
The goal of this interventional study is to evaluate the clinical efficacy of SafeLM™, a video laryngeal mask airway device in paediatric population. The main questions it aims to answer are:

1. To determine the success rate, ease of device insertion, time for insertion, and how well the device seals the airway by measuring the oropharyngeal leak pressure (OPLP) of SafeLM™.
2. To determine the incidence of complication associated with SafeLM™ usage.
3. To study the association of glottic view with success rate and rate of complication.

Participants perioperative clinical data will be collected for data analysis.

DETAILED DESCRIPTION:
Paediatric patients who are scheduled for surgery where supraglottic airway is deemed appropriate will be recruited with written consent. Following preoxygenation, application of standard monitors, and induction of general anaesthesia, an appropriate size of SafeLM™ will be inserted according to manufacturer's recommendation. Cuff will be deflated and flattened prior, with the back of laryngeal mask lubricated. The device will be advanced by sliding the laryngeal mask down the palatopharyngeal curve along the midline in the mouth until the end of the mask reach the hypopharynx cavity and resistance is met, with the process visualised in real time through the video camera. If there is malalignment, correction manoeuvre such as jaw trust, head reposition, or mask redirection will be done. Once the distal end of mask reaches the hypopharyngeal cavity, the cuff is inflated with the recommended volume of air according to the manufacturer recommendation, until adequate cuff seal is achieved. Then, the patient is put on either spontaneous or pressure-controlled mechanical ventilation. Successful placement will be confirmed. If insertion difficulty is encountered and the laryngeal mask is required to be taken out from the oral cavity, insertion can be reattempt with the same or different size of SafeLM™ after adequate preoxygenation, and it will be considered as second attempt. If it remains unsuccessful on the 3rd attempt, SafeLM™ insertion will be abandoned, subsequent management will be decided by the attending anaesthetist. Glottic exposure grades at the end of each attempt is recorded. The time for insertion is measured for each attempt, using a stopwatch, by obtaining the duration in between the moment when the anaesthetist starts holding the SafeLM™ device, until the appearance of 2 complete continuous capnography waveform on the monitor. Following successful SafeLM™ insertion, the camera can be removed, and orogastric tube will be inserted via the gastric port only if there is clinical indication. Subsequently, oropharyngeal leak pressure (OPLP) is measured and recorded by dialing the fresh gas flow rate to 3 L/min and putting the adjusting pressure limiting (APL) valve at 40 cmH2O, in manual ventilation mode. The equilibrium pressure that the pressure gauze pointer settles down at is the OPLP. The anaesthesia is maintained using TIVA or volatile agent as per the anaesthetist's discretion, keeping the MAC at least 1.0 or BIS level at 40-60, whichever is applicable. All the patients will receive IV dexamethasone 0.2 mg/kg and IV granisetron 0.02 mg/kg as post operative nausea vomiting (PONV) prophylaxis. At the end of anaesthesia, anaesthetic agent administration is terminated. If non-depolarising neuromuscular blockade is given during anaesthesia, an appropriate dose of reversal agent will be given according to the depth of neuromuscular blockade based on either clinical signs or nerve stimulation examination, whichever applicable. After the adequate neuromuscular blockade reversal is confirmed, the laryngeal mask can be removed at the awake state or deep plane of anaesthesia. Patient will be monitored in the post-anaesthesia care unit for at least 30 minutes prior sending back to the designated ward for continuation of care.

ELIGIBILITY:
Inclusion criteria

* Patients who are scheduled for a surgery under general anaesthesia where supraglottic airway is deemed appropriate.
* ASA I or II
* Age up to 18 years old
* Body weight of 10 kg and above

Exclusion criteria

* Presence of risk of gastric regurgitation or aspiration
* Recent upper respiratory tract infection within 2 weeks
* Uncontrolled respiratory co-morbidity such as bronchial asthma, chronic lung disease, restrictive lung disease
* Presence of congenital airway abnormalities
* Patient or next of kins refusal in participating this study

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of device placement in percentage | Perioperative
  Percentage of patient experiencing successful insertion of SafeLM™
  The criteria of successful insertion:
  (i) good chest rise during positive pressure ventilation (ii) no significant air leakage (no audible leak on ausculatation, and the ventilator bellow not collapsing (iii) two or more continuous capnography waveforms (iv) able to achieve a minimum expiratory tidal volume of 6ml/kg
  Percetage calculation: number of participants fulfillling successful insertion criteria within 3 insertion attempts divided by total number of participants, multiplied by 100 percents
Oropharyngeal leak pressure (OPLP) in cmH2O | From the time of successful device placement confirmation to the time of determination of OPLP before commencement of surgery
  Oropharyngeal leak pressure (OPLP) is measured and recorded by dialling the fresh gas flow rate to 3 L/min and putting the adjusting pressure limiting (APL) valve at 40 cmH2O, in manual ventilation mode. The equilibrium pressure that the pressure gauze pointer settles down at is the OPLP. The measurement is done after successful device placement confirmation, once OPLP value is obtained, positive pressure ventilation of spontaneous ventilation will resume.
Glottic exposure grades | At the time of completion of device placement procedure, when the distal end of the cuff reaches the hypopharyngeal cavity, resistance is met, and the cuff is inflated with appropriate volume of air as per manufacturer recommendation.
  SaCoVLM™ Glottic exposure grades visualised on the videoscope are recorded for each patient Grade 1: Visualization of the lateral part of the right aryepiglottic fold and part of the laryngeal inlet, and the ventilation was good Grade 2: Visualization of the bilateral aryepiglottic fold and part of laryngeal inlet, and the ventilation was good Grade 3: Visualization of all laryngeal inlet and posterior glottis Grade 4: Visualization of the whole glottis

SECONDARY OUTCOMES:
Insertion time in seconds (s) | Periprocedural
  Time taken for device insertion. The duration in between the moment when the anaesthetist starts holding the SafeLM™ device, until the appearance of 2 complete continuous capnography waveform on the monitor is measured using stopwatch.
The ease of SafeLM™ insertion | Perioperative
  The anaesthetist will rate the ease of SafeLM™ insertion using Likert scale of 1 to 5 (1-Very easy, 2- Easy, 3-Somewhat easy, 4-Difficult, 5-Very difficult). Rating is done at the end of general anesthesia service in the operating theatre.
Anaesthetists' overall satisfactory score | Perioperative
  The anaesthetists' overall satisfactory score will be rated using a scale of 1 to 5 (1-Very dissatisfied, 2-Dissatisfied, 3-Neutral, 4-Satisfied, 5-Very satisfied) Rating is done at the end of general anesthesia service in the operating theatre.
Rate of intraoperative laryngospasm | Intraoperative
  Presence of intra-operative laryngospasm event
Rate of intraoperative bronchospasm | Intraoperative
  Presence of intra-operative bronchospasm event
Rate of intraoperative desaturation event | Intraoperative
  Presence of desaturation event with pulse oximeter value of 90 percent and below
Rate of intraoperative gastric aspiration event | Intraoperative
  Presence of intra-operative gastric aspiration event
Rate of post-extubation gastric aspiration event | Perioperative
  Presence of post-extubation gastric aspiration event from the time of extubation to the time of transfer out from Post anaesthesia care unit (PACU)
Rate of post-extubation sore throat event | Perioperative
  Presence of post-extubation sore throat event from the time of extubation to the time of transfer out from Post anaesthesia care unit (PACU)
Rate of post-extubation finding of blood stain | Perioperative
  Presence of blood stain on the SafeLM™ or oral cavity upon examination during extubation from the time of extubation to the time of transfer out from Post anaesthesia care unit (PACU)
Rate of post-extubation laryngospasm | Perioperative
  Presence of post-extubation laryngospasm event from the time of extubation to the time of transfer out from Post anaesthesia care unit (PACU)
Rate of post-extubation bronchospasm | Perioperative
  Presence of post-extubation bronchospasm event from the time of extubation to the time of transfer out from Post anaesthesia care unit (PACU)

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - University of Malaya, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: Undecided